CLINICAL TRIAL: NCT01978288
Title: Upper Airway Microbial Development During the First Year of Life
Status: Active, not recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Kirsten Kloepfer, Assistant Professor of Pediatric Pulmonology, Allergy and Sleep Medicine, Indiana University
Other Study IDs: 1308055098; K23AI135094 (NIH); 5K12HD068371 (NIH)
Record Dates: First submitted 2013-10-25; First posted 2013-11-07 (Estimated); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal swabs, throat swabs, nasal fluid, blood, and stool specimens will be retained
Oversight: Data Monitoring Committee: Yes | US Export: No

GROUPS / COHORTS (3):
- Cohort 1 Newborns with asthmatic mothers: Infants born to mothers who have diagnosis of Asthma that were enrolled in study from 5/7/14 to 6/1/16.
- Cohort 2 Newborns with asthmatic mothers: Infants born to mothers who have a diagnosis of Asthma with enrollment from June 2, 2016 going forward.
- Cohort 3 Newborns with healthy parents: Infants born to healthy parents without atopy (asthma, eczema, seasonal allergies) from June 2, 2016 going forward.

SUMMARY:
This study tests the hypothesis that an increase in pathogenic bacteria within the infant airway leads to increased airway inflammation, decreased airway function and ultimately airway obstruction throughout the first one to two years of life.

DETAILED DESCRIPTION:
With the prevalence of asthma increasing each decade, our focus has shifted from treatment to understanding the pathogenesis of asthma so we may develop methods of prevention. With the advent of new bacterial detection techniques, we have the opportunity to examine the infant microbiome prior to the development of wheezing and subsequent asthma. Based on our knowledge that certain bacteria are associated with recurrent wheezing, we believe that an increase in pathogenic bacteria alters the airway epithelium resulting in airway inflammation. This chronic inflammation leads to airway obstruction, resulting in recurrent wheezing. By prospectively following children up to two years we have the opportunity to determine if changes seen in early infancy are established early and persist until 2 years of age. In addition, we propose to determine if the microbiome contributes to airway obstruction and episodes of wheezing with respiratory illness. This study tests the hypothesis that an increase in pathogenic bacteria within the infant airway leads to increased airway inflammation, decreased airway function and ultimately airway obstruction throughout the first one to two years of life.

The study has 3 Cohorts:

Cohort 1: Newborns with asthmatic mothers with enrollment from May 7, 2014 to June 1, 2016. Newborns from this cohort meet the below inclusion and exclusion criteria, however they follow a study visit schedule that follows them for 18 months (+/- 6 months).

Cohort 2: Newborns with asthmatic mothers with enrollment from June 2, 2016 going forward. Newborns from this cohort meet the below inclusion and exclusion criteria, however they follow a study visit schedule that follows them for 12 months (+/- 2 months).

Cohort 3: Newborns with healthy parents without atopy from June 2, 2016 going forward. Newborns from this cohort meet the below inclusion and exclusion criteria, however they follow a study visit schedule that follows them for 12 months (+/- 2 months).

Once enrolled, study procedures will consist of: collection of nasal swabs and fluid, stool specimens, and throat swabs, at enrollment visit (first week of life), 3-5 weeks of age (Visit 2), 3-5 months (Visit 3), and 12 months +/- 2 months (Visit 4); blood draw at Visits 3 and 4; spirometry will be performed at Visits 2, 3 and 4: non-sedated infant pulmonary function tests will be conducted at all visits for all cohorts; at Visits 3 and 4, sedated infant pulmonary function tests are optional for Cohorts 1 and 2 only. Finally, surveys will be completed about every two months starting at about two months, then four weeks after Visit 3, and about every 8 weeks until Visit 4, to review infection history, medication (including antibiotics) history and wheezing history.

ELIGIBILITY:
Inclusion Criteria:

1. Moms age 14 and older (will sign Informed Consent Statement (ICS), not an assent)
2. Mother of child enrolled must have a physician diagnosis of asthma or being treated for asthma (for 140 subjects; 40 subjects will be recruited from mothers and fathers without atopy - asthma, eczema, seasonal allergies)
3. Child must be enrolled during first week of life
4. Signed informed consent from parent(s) or legal guardian(s)

Exclusion Criteria:

1. Child has a history of wheezing or underlying lung disease
2. Respiratory complications at birth (airway support higher then nasal cannula)
3. Born earlier then 37 weeks gestation
4. Congenital heart defects (not including Patent Ductus Arteriosus (PDA), hemodynamically insignificant Ventricular Septal Defect (VSD) or Atrial Septal Defect (ASD)
5. Underlying neuromuscular disease
6. Severe upper airway obstruction, sleep apnea, tracheomalacia, or laryngomalacia
7. Hydrocephalus
8. History of seizures
9. History of arrhythmia and baseline oxygenation level <90% on room air
10. Infant is non-viable
11. Severe gastroesophageal reflux
12. Prior chest surgery or structural abnormalities of the lungs or chest wall
13. Has a history of adverse reaction to chloral hydrate
14. Ward of the state
15. Any physical finding(s) that would compromise the safety of the subject or the quality of the study data as determined by the site investigator

Ages: 1 Minute to 1 Week | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants whose mother has asthma; Infants whose parents are without atopy - asthma, eczema, seasonal allergies
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2014-01; Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in airway bacteria diversity during first 12 months of life. | Birth and 12 months (+/- 2 months)
  Will use microbiome diversity measurements to determine if changes in diversity occur over time.

SECONDARY OUTCOMES:
Change in inflammatory markers (IL-4, IL-5 and IL-13) during first 12 months of life. | Birth and 12 months (+/- 2 months)
  c. Determine if the microbiome at age 18 months (+/- 6 months) is associated with decreased lung function and/or increased inflammatory markers.
Change in airway function measurements FEV0.5 during 12 months of life. | Birth and 12 months (+/- 2 months)
  Pulmonary measurements will be obtained. We will look at changes over time in FEV0.5.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Kloepfer, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No